CLINICAL TRIAL: NCT06713811
Title: Evaluation of the Impact of Electronic Monitoring on Patient Compliance in Hematology
Acronym: EMMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Private Hospital of Confluent, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-23-HPC
Record Dates: First submitted 2024-11-25; First posted 2024-12-03 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Hemopathies
Keywords: observance; malignant hemopathies; telemonitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- standard (No Intervention)
- experimental (Experimental)
  Interventions: Other: Telemonitoring

INTERVENTIONS:
Other: Telemonitoring — Cureety is a digital telemonitoring platform specially designed to monitor cancer patients through self-reporting of adverse events. It supports patients and medical teams to complement existing care practices.
  Arms: experimental

SUMMARY:
Management of hemopathies has progressed with the arrival of new drugs such as CAR T-cells (Chimeric Antigen Receptor T-cells), immunotherapy and targeted therapies, while increasing emphasis is being placed on outpatient care.

The emergence of oral therapies has simplified the treatment pathway, but they are not without their undesirable effects, which can sometimes lead to treatment suspension or even discontinuation. These undesirable effects may be related either to the haemopathy (pain, general signs, fatigue, malnutrition, infection, etc.), or to the toxicity of the treatments, or to co-morbidities. It is therefore essential to detect and manage these adverse effects in real time.

In patients treated with oral therapy, poor compliance (<80% of doses taken) can have a direct impact on progression-free survival and sometimes on overall survival (Dashputre et al, Williams et al).

It is therefore imperative for patients to follow prescribed treatments correctly, and for doctors to check for the absence of side-effects that could adversely affect patient safety and quality of life.

Monitoring of these side effects varies from one center to another: it can be "classic", with a call from the patient or GP in the event of an event; it can be telephone-based (AMA-type coordination nurse for Ambulatory Medical Assistance); and finally, it can be electronic via a remote monitoring application.

Monitoring by electronic application has been evaluated in oncology, with a benefit on early detection of side effects or signs of disease progression The human resources and organization of hematology departments are highly heterogeneous, and few studies have been carried out for patients treated long-term (≥ 6 months) with oral therapy.

For these patients, therapeutic compliance is one of the parameters to be assessed, in order to optimize dose-intensity and duration of response.

We propose here to compare two types of follow-up for patients due to start oral therapy: standard follow-up and follow-up by electronic application (Cureety).

ELIGIBILITY:
Inclusion Criteria:

* Follow-up for haemopathy justifying initiation of oral therapy (one or more authorized molecules) for more than 6 months (1st line of treatment or more),
* Intravenous treatment may be associated with it, in accordance with international recommendations (immunotherapy, corticosteroid therapy, other),
* Patient affiliated to a social security scheme,
* Patient having given written consent prior to any specific study procedure.

Exclusion Criteria:

* Oral treatment expected to last < 6 months,
* Cerebral tumor involvement,
* Other active cancer < 3 years, excluding skin, prostate and cervical carcinomas treated by surgery alone,
* Pregnancy or breast-feeding
* Persons deprived of their liberty, under guardianship or curatorship,
* Dementia, mental alteration or psychiatric pathology that could compromise the patient's informed consent and/or compliance with the protocol and trial follow-up,
* Patient unable to undergo protocol monitoring for psychological, social, family or geographical reasons.
* No Internet connection
* No telephone line

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Observance | month 1, month 3, month 6
  Observance will be evaluated by Girerd questionnaire (6 questions : 7 questions with 0 or 1). A score >=3 indicates a poor adhesion, 1-2 is an average adhesion and <6 a good adhesion.

SECONDARY OUTCOMES:
Adverse events | month 1, month 3 and month 6 for control arm ; as they occur for experimental arm
  Adverse events will be reported according to international terminology (CTCAE, Common Terminology Criteria for Adverse Events v5.0), and recorded at each visit for patients in the control arm and by .
Number of unexpected hospitalizations | 6 months
  The number of unexpected hospitalizations will be recorded per arm for the duration of the study
The duration of unexpected hospitalizations | 6 months
  The duration of unexpected hospitalizations will be recorded per arm for the duration of the study
Reason for unexpected hospitalizations | 6 months
  The reason for unexpected hospitalizations will be recorded per arm for the duration of the study

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Clinique de l'Europe, Amiens
  - Clinique de la Baie, Morlaix
  - Hôpital Privé du Confluent, Nantes

IPD SHARING:
Plan to Share IPD: No